CLINICAL TRIAL: NCT03955575
Title: Treatment of Bile Acid Malabsorption With Liraglutide
Acronym: BAM-LIRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Filip Krag Knop (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor-Investigator, Filip Krag Knop, Professor, Consultant Endocrinologist, MD PhD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-18048247
Record Dates: First submitted 2019-03-08; First posted 2019-05-20 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Bile Acid Malabsorption
MeSH Terms: interventions — Liraglutide; Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide/placebo-colesevelam (Active Comparator): Liraglutide as active and colesevelam as placebo
  Interventions: Drug: Liraglutide 6 MG/ML
- Placebo-Liraglutide/colesevelam (Active Comparator): Liraglutide as placebo and colesevelam as placebo
  Interventions: Drug: Colesevelam

INTERVENTIONS:
Drug: Liraglutide 6 MG/ML — Liraglutide as injections.
  Arms: Liraglutide/placebo-colesevelam
Drug: Colesevelam — 3 x 625 miligram 2 times a day.
  Arms: Placebo-Liraglutide/colesevelam

SUMMARY:
Comparing the effect of Liraglutide on bile acid malabsorption, with colesevelam

DETAILED DESCRIPTION:
The overall objective of the present study is to provide proof of concept that treatment with the GLP-1 receptor agonist liraglutide is efficacious (as assessed by symptom relief, i.e. response to treatment) and safe (as assessed by adverse effects) in the management of BAM and that it improves bile acid reabsorption (as assessed by SeHCAT) in these patients.

ELIGIBILITY:
Inclusion Criteria:

* • Caucasian ethnicity

  * SeHCAT-verified moderate (5-10% bile acid retention after 7 days) or severe BAM (<5% retention)
  * Normal haemoglobin (for men 8.3-10.5 mmol/L; for women 7.3-9.5 mmol/L)
  * Age above 18 years and below 75 years
  * Informed and written consent
  * BMI >18,5 kg/m2 and <40 kg/m2
  * Glycated haemoglobin (HbA1c) <48 mmol/mol

Exclusion Criteria:

* • History of or present hepatobiliary disorder (except for non-alcoholic steatotic liver disease) and/or alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >3 times upper limit of normal) or history of hepatobiliary disorder

  * Gastrointestinal disease (except for BAM), previous intestinal resection or any major intra-abdomial surgery
  * Diabetes mellitus
  * Nephropathy with eGFR < 60 mL/min/1.73m2
  * Treatment with medicine that cannot be paused for 12 hours
  * Hypothyroidism or hyperthyroidism, if not well regulated.
  * Treatment with oral anticoagulants
  * Active or recent malignant disease
  * Any treatment or condition requiring acute or sub-acute medical or surgical intervention
  * Females of child-bearing potential who is pregnant (tested before entering the study), breastfeeding or intend to become pregnant or is not using adequate contraceptive methods, which includes Intrauterine Device (IUD), birth control pills, sexual abstinence or living in a relationship with a sterile partner.
  * Known or suspected hypersensitivity to trial products or related products
  * Any condition considered incompatible with participation by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in stool fequency | 7 weeks
  Contestants will use a questionaire, which will be filled out three times during the 7 weeks periode

SECONDARY OUTCOMES:
Total symptoms score, quality of life scores, and biomarker. | 7 weeks
  Total symptoms score, quality of life scores, and biomarker values will be analysed using a constrained linear mixed model with inherent baseline adjustment and with an unstructured covariance pattern. Changes since baseline within and between groups will be reported with 95% confidence intervals.
Change in SeHCAT | 7 weeks
  Three SeHCAT scans will be made, and the difference will be evaluated
Proportions of patients tolerating the treatment and proportion of patients experiencing remission of BAM related diarrhoea | 7 weeks
  Proportions of patients tolerating the treatment and proportion of patients experiencing remission of BAM related diarrhoea within each group will be reported with exact binomial confidence intervals and compared between groups using risk differences and Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD PhD, Principal Investigator — filip.krag.knop.01@regionh.dk
Locations (1):
- Gentofte Hospital, Hellerup, Regionh, Denmark

IPD SHARING:
Plan to Share IPD: No